CLINICAL TRIAL: NCT02572947
Title: An Interventional, One-arm, Open Label Pilot Study to Assess the Feasibility of Dolutegravir Monotherapy in Virologically Suppressed Patients on Conventional Triple Antiretroviral Therapy of Dolutegravir Plus Two Nucleoside Reverse Transcriptase Inhibitors
Brief Title: A Pilot Study of MONOtherapy of DOlutegravir in HIV-1 Virologically Suppressed Patients
Acronym: MONODO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Calmy Alexandra (Other)
Responsible Party: Sponsor-Investigator, Calmy Alexandra, Médecin adjointe agrégée, HIV Unit director, Infectious Diseases Division, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRD-13-2015-I
Record Dates: First submitted 2015-10-07; First posted 2015-10-09 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Human Immunodeficiency Virus; Dolutegravir; Monotherapy; Treatment Efficacy
Keywords: Dolutegravir; HIV infection; Anti-Retroviral Agents; HIV Integrase Inhibitors; Integrase Inhibitors; Pharmacologic Actions; Therapeutic Uses
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dolutegravir monotherapy (Experimental): 10 patients will be simplified to monotherapy of dolutegravir tablet 50mg once daily for 24 weeks
  Interventions: Drug: Dolutegravir

INTERVENTIONS:
Drug: Dolutegravir

SUMMARY:
Current HIV treatment guidelines recommend a combination of drugs for the maintenance of antiretroviral therapy (ART). Simplification is considered critical to further scale-up of treatment, to support retention in care and to reduce costs. Dolutegravir is a once daily integrase inhibitor that shows very good tolerability, efficacy, and distinctive resistance profile. The researchers aim at investigating the feasibility of dolutegravir monotherapy in maintenance therapy. Briefly, 10 virologically suppressed patients for at least six months on conventional triple ART of dolutegravir plus two nucleoside reverse transcriptase inhibitors (NRTIs) will be switched to dolutegravir monotherapy for 24 weeks. The primary endpoint is the number of patients completing 24 weeks of dolutegravir monotherapy without experiencing virological failure.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection;
* Patient included in the Swiss HIV Cohort Study (SHCS);
* ≥ 18 years of age;
* Virologically suppressed for at least 24 months on first line triple ART (changes for toxicity permitted) with at least 4 HIV-1 RNA measurements in plasma <50 copies/ml;
* No history of previous failure on ART;
* No documented antiretroviral drugs resistance;
* No co-infection with Hepatitis B or C virus;
* Effective contraception in women;
* Willing to provide CSF and semen samples;
* Written informed consent

Exclusion Criteria:

* HIV-2 infection;
* Renal dysfunction (creatinine clearance <50ml/min);
* aspartate transaminase or alanine aminotransferase >5x upper limit normal;
* Concomitant use of carbamazepine, oxcarbazepine, phenytoin, phenobarbital, St John's wort, rifampicin or metformin;
* Previous AIDS defining conditions or active malignancy in the past five years;
* Positive HIV viral load in CSF at baseline;
* Known or suspected non-compliance;
* Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-06; Primary Completion 2017-06 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Number of patients without virological failure defined as plasma HIV-1 RNA ≥ 200 copies/ml on two consecutive measurements or positive HIV-1 RNA level in cerebrospinal fluid (CSF) at week 24 or before | week 24

SECONDARY OUTCOMES:
Quantification of the HIV-1 DNA reservoir in peripheral blood monocyte cells at baseline and week 24 | week 24
Emergence of genotypic resistance in plasma HIV-1 RNA in case of virological failure | week 24
Quantification HIV-1 RNA levels in the CSF and semen at baseline and week 24 | week 24
  Lumbar puncture is optional at baseline
Change from baseline CD4 cell count from baseline at week 24 | week 24
Adherence to medication at weeks 4, 8, 12, 16, 20, 24 | week 24
  Number of participants with suboptimal adherence defined as more than 3 pills (10%) remaining from previous monthly visit OR missed more than one dose in a row OR missed dose more than once every two weeks
Lipidic profile changes from baseline at week 24 | week 24
Body fat composition as measured by dual energy x-ray absorptiometry (DXA) scan at baseline and week 24 | week 24
Change in bone mineral density from baseline to week 24 | week 24
  Number of patients with normal bone density, osteopenia or osteoporosis as defined by DXA scans results

OTHER OUTCOMES:
Change in immune activation from baseline to week 24 measured by highly sensitive C-reactive protein (mg/l) | week 24
Change in immune activation from baseline to week 24 measured by cytokines (pg/ml) | week 24
Change in immune activation from baseline to week 24 measured by d-dimers (microg/l) | week 24

CONTACTS AND LOCATIONS:
Overall Officials: Delphine Sculier, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hospitals of Geneva, HIV unit, Geneva, Switzerland